CLINICAL TRIAL: NCT03755583
Title: Effect of Exclusive Enteral Nutrition on Disease Process, Nutritional Status and Intestinal Microbiota for Chinese Children With Crohn's Disease
Brief Title: Effect of Exclusive Enteral Nutrition on Disease Process, Nutritional Status and Gastrointestinal Microbiota for Chinese Children With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBD-EEN-microbiota
Record Dates: First submitted 2018-11-18; First posted 2018-11-28 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Crohn Disease; Enteral Nutrition; Gastrointestinal Microbiome
Keywords: Exclusive enteral nutrition
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEN group (Other): Received exclusive enteral nutrition after enrollment.
  Interventions: Dietary Supplement: Exclusive Enteral Nutrition

INTERVENTIONS:
Dietary Supplement: Exclusive Enteral Nutrition — a complete liquid diet of formula for 8 weeks were adminstered in Crohn's Diseas patients ,Nutritional intake was based on the child's estimated energy requirements, no regular table food during 8 weeks treament.

SUMMARY:
Inflammatory bowel diseases (IBD) are chronic inflammatory diseases. It is believed that the inflammation results from sustained abnormal immune response towards altered or pathogenic microbiota in genetically susceptible hosts. Malnutrition is common in IBD, especially in pediatric Crohn's disease(CD). Exclusive enteral nutrion(EEN) has been shown to improve nutritional status and inflammatory markers in pediatric CD. But there is limited data about the effect of EEN on Chinese children with CD. In this study, investigators focused on disease process,nutritional status and gut microbiome of Chinese children with newly-diagnosed CD after EEN treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric CD patients who were newly diagnosed and being treated with EEN at the Children's Hospital of Fudan University

Exclusion Criteria:

* (1) patients who were administered corticosteroids, immunosuppressive drugs, or biological agents prior to the study; (2) patients who could not finish the daily prescribed volume of formula for any reason; (3) patients who could not attend consecutive follow-up sessions; (4) patients who had received antibiotics or probiotics within 1.5 months prior to the study; and (5) patients who had been given corticosteroids, immunosuppressive drugs, biological agents, antibiotics, or probiotics during the EEN process.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
5-item gut microbiota measure | 0, 2, 6, 8, 12 weeks post-EEN
  the change of gut microbiota during EEN and after the end of EEN
2-item Simple Endoscopic Score for CD (SES-CD) | 0, 8, weeks post-EEN
  According to the SES-CD, at the end of EEN, the patients whose SES-CD scores were ≤4 were classified into the remission group (CD-RE), other patients whose SES-CD scores were >4 were classified into the non-remission group (CD-NRE)

SECONDARY OUTCOMES:
5-item weighted Paediatric Crohn's disease activity index measure(wPCDAI) | 0, 2, 6, 8, 12 weeks post-EEN
  wPCDAI scoret included 8 items (Abdominal pain, Patient functioning, Stools, ESR, Albumin, Weight, Perirectal disease, Extraintestinal manifestations ).
2-item 25-hydroxyvitamin D3 measure (25-OH VITD3) | 0,8 weeks post-EEN
  the level of 25-OH VITD3 in 8 weeks post-EEN is higher than 0 week represents a better outcome
5-item weight measure | 0, 2, 6, 8, 12 weeks post-EEN
5-item height measure | 0, 2, 6, 8, 12 weeks post-EEN
5-item Fecal Calprotectin | 0, 2, 6, 8, 12 weeks post-EEN
2-item Insulin-like growth factor-1 | 0, 8 weeks post-EEN
2-item Calcium, vitamin | 0, 8 weeks post-EEN

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided